CLINICAL TRIAL: NCT04680078
Title: A Comparison Between Placement of Three Interrupted Sutures After Triangular Three-snip Punctoplasty vs Conventional Triangular Three-snip Punctoplasty for Treatment of Lower Punctal Stenosis
Brief Title: Placement of Three Interrupted Sutures After Triangular Three-snip Punctoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Abdulhady, Resident doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MenoufiaU112019
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Epiphora
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placement of three interrupted sutures after Triangular Three-snip Punctoplasty of the lower punctum (Active Comparator): After instillation of topical benoxinate hydrochloride 0.4%, subconjunctival injection of 2% lidocaine was done beneath the lower punctum, then Nettleship dilator was used to dilate the punctum. A single blade of a small Westcott spring scissor or Vannus scissor is placed within the ampulla of the lacrimal canaliculus, with the remaining blade placed on the conjunctival surface of the posterior aspect of the eyelid. The first vertical snip is made at the vertical canaliculus. The second vertical snip is made from the edge of the first snip to create a flap. The final horizontal snip was made at the base. The triangular flap is removed and three sutures are placed, in an interrupted manner, at the posterior wall of the ampulla using 10-0 nylon. Hemostasis was done by compression with a cotton tip for one minute until bleeding stop. The sutures are removed 1 week after the surgery.
  Interventions: Procedure: Placement of three interrupted sutures after Triangular Three-snip Punctoplasty of the lower punctum
- Conventional Triangular Three-snip Punctoplasty of the lower punctum (Active Comparator): After instillation of topical benoxinate hydrochloride 0.4%, subconjunctival injection of 2% lidocaine was done beneath the lower punctum, then Nettleship dilator was used to dilate the punctum. A single blade of a small Westcott spring scissor or Vannus scissor is placed within the ampulla of the lacrimal canaliculus, with the remaining blade placed on the conjunctival surface of the posterior aspect of the eyelid. The first vertical snip is made at the vertical canaliculus. The second vertical snip is made from the edge of the first snip to create a flap. The final horizontal snip was made at the base. Hemostasis was done by compression with a cotton tip for one minute until bleeding stop.
  Interventions: Procedure: Conventional Triangular Three-snip Punctoplasty of the lower punctum

INTERVENTIONS:
Procedure: Placement of three interrupted sutures after Triangular Three-snip Punctoplasty of the lower punctum — A Nettelship dilator is used to enlarge the stenotic lacrimal punctum. A single blade of a small Westcott spring scissor or Vannus scissor is placed within the ampulla of the lacrimal canaliculus, with the remaining blade placed on the conjunctival surface of the posterior aspect of the eyelid. The first vertical snip is made at the vertical canaliculus. The second vertical snip is made from the edge of the first snip to create a flap. The final horizontal snip was made at the base. The triangular flap is removed and three sutures are placed, in an interrupted manner, at the posterior wall of the ampulla using 10-0 nylon. The sutures are removed 1 week after the surgery.
  Arms: Placement of three interrupted sutures after Triangular Three-snip Punctoplasty of the lower punctum
Procedure: Conventional Triangular Three-snip Punctoplasty of the lower punctum — A Nettelship dilator is used to enlarge the stenotic lacrimal punctum. A single blade of a small Westcott spring scissor or Vannus scissor is placed within the ampulla of the lacrimal canaliculus, with the remaining blade placed on the conjunctival surface of the posterior aspect of the eyelid. The first vertical snip is made at the vertical canaliculus. The second vertical snip is made from the edge of the first snip to create a flap. The final horizontal snip was made at the base. The triangular flap is then removed .
  Arms: Conventional Triangular Three-snip Punctoplasty of the lower punctum

SUMMARY:
a prospective randomized study conducted upon 40 eyes of 24 patients with lower punctual stenosis (grade 1 or 2 according to Kashkouli scale) attending at Menoufia University hospitals and Kafr Elsheikh ophthalmic eye center. The upper punctum and canaliculus were patent. All patients were complaining of epiphora and had a thorough ophthalmological examination including dye disappearance test, and slit-lamp examination. A Nettelship dilator is used to enlarge the stenotic lacrimal punctum. A single blade of a small Westcott spring scissor or Vannus scissor is placed within the ampulla of the lacrimal canaliculus, with the remaining blade placed on the conjunctival surface of the posterior aspect of the eyelid. The first vertical snip is made at the vertical canaliculus. The second vertical snip is made from the edge of the first snip to create a flap. The final horizontal snip was made at the base. The triangular flap is removed and three sutures are placed, in an interrupted manner, at the posterior wall of the ampulla using 10-0 nylon. The sutures are removed 1 week after the surgery. Topical moxifloxacin 0.5% eye drops and fluorometholone 0.1% eye drops were used four times daily for one week.Patients were then followed up for 6 months after the surgery.

DETAILED DESCRIPTION:
This is a prospective non-randomized study which includes 40 eyelids of 24 patients with acquired lower punctal stenosis grade 1 or grade 2 according to Kashkouli scale attending at Menoufia University hospitals and Kafr Elsheikh ophthalmic eye center in the period from January 2019 to June 2020. Ethics approval from the institutional review board was obtained, and a written informed consent was taken from every patient according to the Declaration of Helsinki.

A full history and examination were done for patients for evaluation of proximal lacrimal drainage system and exclusion of other causes of epiphora rather than punctal stenosis, Inspection of face and periorbital region for position of the eyelids and puncta, Gross nasal deformity, Facial symmetry, presence of any swelling or fistula in the lacrimal sac area , palpation of lacrimal sac for regurge test , slitlamp examination of lid margin for coaptation with the globe , blepharitis or rubbing lashes , skin for laceration or eczema , conjunctiva for papillae , follicles, hyperemia or discharge , cornea for punctate keratitis, filaments or abrasions , lower Tear meniscus height (TMH) using a 1 mm slit beam , punctal orifices position, shape , grading of stenosis according to Kashkouli et al.

Fluorescein dye disappearance test (FDDT) where the fluorescence of the tear meniscus was observed with the help of cobalt-blue filter. FDDT was graded according to Ozgur et al., scale according the time of dye clearance.

Diagnostic probing and syringing were done to ensure anatomically patent nasolacrimal system and to detect any obstruction distal to the punctum.

Patients were examined for results in visits at one week, 1month, 3 months and 6 months.

Satisfactory surgical outcome was defined as postoperative patent lower eyelid punctum and improved Epiphora and FDDT grade at 6 months after surgery.

Surgical procedure

Surgery was performed using an operating microscope under local anaesthesia. We transconjunctivally infiltrate 2% (w/v) lidocaine (with epinephrine in a 1:100,000 weight ratio) from the posterior aspect of the eyelid into the region of the lacrimal canaliculus and punctum.A Nettelship dilator is used to enlarge the stenotic lacrimal punctum. A single blade of a small Westcott spring scissor or Vannus scissor is placed within the ampulla of the lacrimal canaliculus, with the remaining blade placed on the conjunctival surface of the posterior aspect of the eyelid. The first vertical snip is made at the vertical canaliculus. The second vertical snip is made from the edge of the first snip to create a flap. The final horizontal snip was made at the base. The triangular flap is removed and three sutures are placed, in an interrupted manner, at the posterior wall of the ampulla using 10-0 nylon. The sutures are removed 1 week after the surgery. Topical moxifloxacin 0.5% eye drops and fluorometholone 0.1% eye drops were used four times daily for one week.Patients were then followed up in 1 week , 1 month , 3 months , 6 months period.

ELIGIBILITY:
Inclusion Criteria:

* primary acquired lower punctal stenosis grade 1 or 2 according to Kashkouli et al. , patent upper punctum and both canaliculi as well as patent nasolacrimal duct , normal lower eyelid margin position

Exclusion Criteria:

* Patients with Congenital punctal stenosis, Acute conjunctival allergic punctal stenosis, Punctal stenosis associated with radiotherapy, Lid malposition, Canalicular, lacrimal sac and nasolacrimal duct obstruction revealed after syringing , Previous eyelid or lacrimal drainage system surgery, Blepharitis and ocular surface disorders, Patients with dry eye were excluded.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-23 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement of epiphora by Munk score | 6 months
  Measurement of improvement of epiphora by use of Munk score as follow :
  Grade 0 : No Epiphora. Grade 1 : Occasional epiphora requiring drying or dabbing less than twice a day.
  Grade 2 : Epiphora requiring dabbing two to four times per day. Grade 3 : Epiphora requiring dabbing five to ten times per day. Grade 4 : Epiphora requiring dabbing more than ten times daily or constant tearing.
Degree of improvement of lacrimal drainage by Dye disappearance test | 6 months
  Performed by putting a drop of 2% fluorescein sodium in the conjunctival sac followed by assessment after 5 minutes of the remaining dye in the tear meniscus. Results were graded according to the following scale
  Grade 1 : <3 minutes Grade 2 : 3-5 minutes Grade 3 : >5 minutes
Slit lamp assesment of the state of the lower punctum | 6 months
  Slit lamp examination of the lower punctum and its grading according to Kashkouli scale as follows:
  Grade 0 : No punctum (agenesis) Grade 1 : Papilla is covered with a membrane (difficult to recognize) Grade 2 : Less than normal size, but recognizable Grade 3 : Normal Grade 4 : Small slit (<2 mm) Grade 5 : Large slit (≥2 mm)

CONTACTS AND LOCATIONS:
Overall Officials: sameh s mandour, MD, Principal Investigator — Menoufia University
Locations (1):
- MenoufiaU, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No